CLINICAL TRIAL: NCT01573208
Title: Prospective Cohort of FIRST TKA With Custom Guides
Brief Title: Custom Guides for Total Knee Arthroplasty (TKA)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Brigitte Jolles, MD, Prof., University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO 278/10
Record Dates: First submitted 2012-03-22; First posted 2012-04-09 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

ARMS (1):
- Register (Experimental): Register
  Interventions: Device: Custom guides

INTERVENTIONS:
Device: Custom guides — Symbios custom guides for TKA

SUMMARY:
The goal of the study is to know if the reconstruction of the lower limb mechanical axis and the patient knee function is improved after Total Knee Arthroplasty (TKA) using patient specific instruments.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a TKA
* Informed signed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-11 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Changes in mechanical axis of the lower limb | Pre-operatively (up to 3 months);6months
  Mechanical axis of the lower limb as defined by the X-Ray evaluation form of the Knee Society Score
Changes in gait | Pre-operatively (up to 3 months); 6 months
  Spatio temporal parameters of the gait

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV - Site HO, Lausanne, CH, Switzerland